CLINICAL TRIAL: NCT03811405
Title: Physiology, Imaging and Modeling of Deep Brain Stimulation for Essential Tremor
Brief Title: Physiology, Imaging and Modeling of Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802397 -N -A; OCR19607 (Other: UF OnCore); 5R25NS108939-04 (NIH); MEDTRONIC INC (Other: AGR00011004)
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Essential Tremor; Parkinson Disease; Dystonia
Keywords: Deep Brain Stimulation (DBS); ventralis intermedius nucleus (VIN); implantable pulse generator (IPG); Diffusion Tensor Imaging (DTI)
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Dystonia

STUDY DESIGN:
Intervention Model Description: Patients with chronically implanted DBS devices for ET who experience progressive worsening of tremor symptoms over time.
Masking Description: Each of the 3 interventions will be videotaped for blinded motor score assessment by an independent rater.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with Essential Tremor (Experimental): Patients with chronically implanted DBS devices for ET who experience progressive worsening of tremor symptoms over time. The DBS implantable pulse generator (IPG) will be loaded with a temporary custom firmware to allow implementation of active biphasic pulse stimulation. The following random conditions will be applied: (1) Home Settings; (2) VIN Biphasic; (3) Stimulator Off. A 30-minute washout period will be applied between each of the random conditions. Therefore, each patient will serve as their own control.
  Interventions: Device: Active biphasic pulse stimulation---Home Settings; Device: Active biphasic pulse stimulation---VIN Biphasic; Device: Active biphasic pulse stimulation---Stimulator Off

INTERVENTIONS:
Device: Active biphasic pulse stimulation---Home Settings — During this visit, the DBS implantable pulse generator (IPG) will be loaded with a temporary custom firmware to allow implementation of active biphasic pulse stimulation.
Device: Active biphasic pulse stimulation---VIN Biphasic — During this visit, the DBS implantable pulse generator (IPG) will be loaded with a temporary custom firmware to allow implementation of active biphasic pulse stimulation.
Device: Active biphasic pulse stimulation---Stimulator Off — During this visit, the DBS implantable pulse generator (IPG) will be loaded with a temporary custom firmware to allow implementation of active biphasic pulse stimulation.

SUMMARY:
This project aims to investigate novel ways to deliver brain stimulation to Essential Tremor (ET) patients by introducing software changes to their existing devices. The study team aims to investigate safety and efficacy of these new stimulation parameters in patients with ET.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is a neuromodulatory therapy that is effective in a subset of well selected essential tremor (ET) patients. However, as many as 1/5 of patients may initially improve, but then steadily worsen following the operation. The investigators developed a technique to study a variety of alternative stimulation methods without the use of an invasive repeat surgical intervention.

The electrophysiological effects of non-conventional DBS differ from traditional DBS, however the physiological differences in the setting of human tremor remain largely unknown. This study plans to explore gaps in knowledge of neuromodulation and will collect and contribute essential information to the underlying mechanism of action of DBS. The hypothesis of this project centers around active biphasic stimulation providing a wider therapeutic window and a lower adverse event profile as compared to conventional DBS.

ELIGIBILITY:
Inclusion Criteria:

* Existing unilateral or bilateral VIN DBS for ET, non-demented (MMSE>24), and must have a documented suboptimal tremor suppression on two successive visits (compared to the baseline post-operative improvement at 6 months following ET DBS surgery). For bilateral cases, the most affected tremor side will be studied.

Exclusion Criteria:

* No diagnosis of Essential Tremor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Volume of tissue activated from stimulation with ET DBS | up to 24 hours
  The study team will use computer simulation and virtual reconstruction of the brain from pre-operative MRI data to calculate the volume of tissue activated (VTA) from the novel stimulation patterns. The investigators will assess the feasibility of the patterns to address the worsening of ET that may occur in 20% or more of the ET population.
Baseline DBS settings versus active biphasic pulse DBS settings | up to 1 hour
  The investigators will compare the degree of tremor suppression from the most optimal DBS settings that can be obtained via traditional programming methods versus active biphasic DBS. The degree of tremor will be quantified by multiple clinical metrics including the Fahn-Tolosa-Marin Tremor Rating Scale and Kinesia ONE® accelerometer system.

SECONDARY OUTCOMES:
The Fahn-Tolosa-Marin Tremor Rating Scale | up to 15 minutes
  Essential tremor severity will be assessed by the clinically validated Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS). It is a 0 to 4 scale (0 = no tremor; 4 = severe amplitude of tremor) of 9 different parts of the body. The FTMTRS will be assessed for the various DBS settings.
Tremor motor physiology | up to 15 minutes
  Essential tremor motor physiology will be recorded by the Kinesia ONE accelerometer system. THe Kinesia ONE system is a wireless wearable motion sensor unit and portable transducer that translates the degree of movement into a standardized scale. Tremor physiology will be assessed for the various DBS settings.
Gait impairment | up to 15 minutes
  Essential tremor's effect on gait will be assessed by the GAITRite system. Patients will walk along a GAITRite floor mat to have the various gait parameters such as step time, cycle time, step length, stride length, etc measured. Gait parameters will be assessed on the various DBS settings.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua K Wong, MD, Principal Investigator — Univeristy of Florida
Locations (2):
- United States (2):
  - UF Health at the University of Florida, Gainesville, Florida
  - McKnight Brain Institute--Fixel Center for Neurological Diseases, Gainesville, Florida